CLINICAL TRIAL: NCT00379275
Title: Ocular and Immuno-Genetic Manifestations of Sarcoidosis
Brief Title: Eye and Immunogenetic Features of Sarcoidosis
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060239; 06-EI-0239
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Sarcoidosis; Uveitis
Keywords: Sarcoidosis; Uveitis; Pulmonary Sarcoidosis; HLA-Typing; Cytokines; Serum Markers
MeSH Terms: conditions — Sarcoidosis; Uveitis; Sarcoidosis, Pulmonary

SUMMARY:
This study will evaluate patients with sarcoidosis to understand how the disease affects the body. Sarcoidosis is a disease that results from inflammation of body tissues. The lungs, lymph nodes in the chest, skin and eyes are most commonly affected. As the disease progresses, small lumps, or granulomas, appear in the affected tissues. In most cases, the granulomas clear up, but in cases where they do not heal and disappear, the tissues tend to remain inflamed. Eye inflammation (uveitis) associated with sarcoidosis can cause various eye diseases, sometimes leading to blindness. This study will examine the clinical, immunological and genetic features of ocular sarcoidosis.

Patients 6 years of age and older with sarcoidosis may be eligible for this study. Candidates are screened with the following procedures:

* Completion of a questionnaire with medical, social and demographic information
* Blood draw for laboratory tests
* Complete eye examination, including measurement of eye pressure and dilation of the pupils to examine the back of the eye. Fluorescein angiography may be done. This test involves injecting a dye into a vein in the arm. The dye travels to the blood vessels in the eyes. A camera flashes a blue light into the eye and takes pictures of the retina that show whether the dye has leaked from the blood vessels into the retina. Other photographs of the eye may also be taken using a special camera.

Participants are followed in conjunction with their local eye doctor as required by the status of their disease. Patients whose disease is stable are seen for an initial examination and followed every 12 months for 3 years.

DETAILED DESCRIPTION:
BACKGROUND

Sarcoidosis is a multi-systemic granulomatous disease. The lungs, thoracic lymph nodes, the skin and the eyes are the most commonly affected organs. Most patients with sarcoidosis present with respiratory symptoms. Sarcoid uveitis is usually suspected when ocular inflammation is found in conjunction with suggestive serological and radiological studies. Currently, the diagnosis of sarcoidosis requires the demonstration of non-caseating granulomas on biopsy; but even this is not always diagnostic; more sensitive and specific noninvasive tools are needed.

Ophthalmic involvement has been reported in as many as 40% of patients with sarcoidosis, but most series report ophthalmic findings in approximately 25% of patients who develop chronic, systemic sarcoidosis. Uveitis associated with sarcoidosis can be very diverse, including: acute non-granulomatous or chronic granulomatous iridocyclitis, vitritis, retinal vasculitis, choroiditis with choroidal granulomas and papillitis secondary to optic nerve granulomas; and it can cause ocular morbidity due to a high incidence of glaucoma and cataracts. Other ophthalmic findings include lacrimal gland enlargement, secondary Sjogren's disease, scleritis, orbital gland involvement, secondary proliferative retinopathy, subretinal neovascularization, and optic neuropathy.

To better evaluate and diagnose patients, we also need to improve our ability to predict susceptibility and prognosis, especially among African-Americans. Current epidemiologic studies of sarcoidosis indicate that in the United States, African Americans have about a threefold higher age-adjusted annual incidence, 35.5/100,000, compared with Caucasians, 10.9/100,000. In addition, African Americans with chronic sarcoidosis are more likely to develop ocular manifestations than whites. The study of ocular sarcoidosis is important because it is a leading inflammatory cause of blindness and ocular morbidity. In large surveys of patients with uveitis, approximately 5% of patients were found to have ocular sarcoidosis, and approximately 10% of these patients become blind in at least one eye.

AIMS:

AIM 1: CLINICAL ANALYSIS:

Documentation of:

1. Clinical features of sarcoidosis associated uveitis
2. Chronological association of ocular disease to histopathologic diagnosis of sarcoidos
3. Family history of sarcoidosis
4. Previous therapies and response
5. Ocular status compared with systemic disease status, current and historical Environmental exposure history

AIM 2: IMMUNOLOGICAL ANALYSIS:

One of the goals of this study is to determine the diagnostically important cytokines in biopsy-proven ocular sarcoidosis.

The chemokine profile of the Peripheral Blood Mononuclear Cells and Broncho-Alveolar Lavage Fluid (BALF) of pulmonary sarcoidosis patients has been reported and many cytokines have been implicated in the pathogenesis of this disease.

1. Serum Level for

   A. TNF alpha

   B. MIP-1 alpha

   C. IL-8

   D. IL-2

   E. TGF Beta

   F. INF gamma
2. Immunophenotyping of whole blood cells and BALF by flow cytometry

   Focus on:

   A. T cell sub-typing (examples: CD4, CD8)

   B. NK cell sub-typing (examples:CD56, KIR)
3. TLRs sub-typing

AIM 3: GENETIC ANALYSIS:

Serum analysis for HLA Class I and II typing

A cohort of 100 patients with biopsy-proven sarcoidosis will be recruited from the Uveitis and Ocular Immunology Clinic at the National Eye Institute and the Pulmonary Clinic at the National Heart Lung and Blood Institute.

FUTURE AIMS:

We aim to characterize the TLR activation profile in patients with ocular sarcoidosis, and compare them to patients with pulmonary sarcoidosis and normal volunteers. Using this immuno-genetic classification scheme, in conjunction with HLA typing, we hope to develop novel diagnostic and/or prognostic criteria for sarcoidosis. In addition, the TLR activation profile may allow risk stratification for different sarcoidosis phenotypes.

METHODS:

A cohort of 100 patients with biopsy-proven sarcoidosis will be recruited from the Uveitis and Ocular Immunology Clinic at the National Eye Institute and the Pulmonary Clinic at the National Heart Lung and Blood Institute. After obtaining informed consent, the patients will be invited to participate in the study. After appropriate enrollment, they will undergo the following

1. Completion of a questionnaire, with medical, social and demographic data
2. A complete ophthalmologic examination
3. Baseline serologic analysis
4. Baseline serum analysis for immunologic analysis
5. HLA-Typing
6. Patients who are quiescent will be seen at baseline with a second visit at 1 year
7. Patients who are active will be treated appropriately, by their referring ophthalmologist or on a treatment protocol at the National Eye Institute

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participants must be at least 6 years old
  2. Participants must have biopsy-proven sarcoidosis
  3. Participant must be able to consent to participating in the protocol
  4. For minors, consent by an adult will be necessary

EXCLUSION CRITERIA:

We will exclude participants who are unable or unwilling to give blood at the designated times in the protocol

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2006-09-18; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jabs DA, Johns CJ. Ocular involvement in chronic sarcoidosis. Am J Ophthalmol. 1986 Sep 15;102(3):297-301. doi: 10.1016/0002-9394(86)90001-2. PMID 3752193